CLINICAL TRIAL: NCT03179189
Title: Investigation of The Prevalence of Sepsis in Adults in Multicenter Intensive Care Unıts in Turkey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilhan bahar, MD,Critical care, Izmir Ataturk Training and Research Hospital
Other Study IDs: 2017/77
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pathophysiology and treatment of sepsis disease are still not fully known. International guides often refer to the studies done in the developed countries and suggest some treatments. The infrastructure of the developing countries is quite different. For this reason, it is not exactly scientific how much these proposals are reflected in patient treatment. In our study, We will try to reveal the treatment of sepsis.

DETAILED DESCRIPTION:
Sepsis is a clinical syndrome that has physiologic, biologic, and biochemical abnormalities caused by a dysregulated inflammatory response to infection. Sepsis and the inflammatory response that ensues can lead to multiple organ dysfunction syndrome and death. In the late 1970s, it was estimated that 164,000 cases of sepsis occurred in the United States (US) each year. Since then, rates of sepsis in the US and elsewhere have dramatically increased as supported by the following studies, although many of these are derived from academic institutions. The increased rate of sepsis is thought to be a consequence of advancing age, immunosuppression, and multidrug-resistant infection. It is also likely to be due to the increased detection of early sepsis from aggressive sepsis education and awareness campaigns, although this hypothesis is unproven. Guidelines should focus on pre-hospital assessment and triage. Indeed, respiratory infections represented the most common cause of sepsis in that cohort, and postoperative infections were another important part of the problem. Whether these conditions apply to patients with shock in low-income and middle-income countries (LMIC) is unknown, but the incidence of community-acquired infections would be higher, with a greater prevalence of gastroenteritis, septic abortion, and skin and soft tissue infections as causes of septic shock. The bacteriology of bloodstream infections across LMICs varies substantially depending on regional and population characteristics. In a meta-analysis of 19 prospective studies on community-acquired bacteraemia in Africa, the most common organisms isolated were Salmonella spp (predominantly non-typhi), Streptococcus pneumoniae, and Gram-negative organisms such as Escherichia coli.11 Among cases for which mortality data were recorded, patients with bloodstream infections had an average mortality of 21.5%. Although data are lacking, appropriate antibiotic treatment for these infections on the basis of bacterial resistance patterns will ultimately depend on the ecological pressures resulting from local antibiotic availability and patterns of use.

We aimed to evaluate the approach to sepsis in Turkey as a multi-centered study.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old over

Exclusion Criteria:

* Non-life expectant Those who live longer than 24 hours not that consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and over
Study Population: propective chort
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
sepsis mortality | 90 day

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk education research izmir, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided